CLINICAL TRIAL: NCT03454815
Title: Effect of Apical Patency on Success of Primary Non-surgical Root Canal Treatment in Non Vital Teeth - a Prospective Study
Brief Title: Effect of Apical Patency on Success of Root Canal Treatment in Non Vital Teeth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Mayank Arora Thesis
Record Dates: First submitted 2018-02-19; First posted 2018-03-06 (Actual); Last update posted 2018-03-06 (Actual); Status verified 2018-03

CONDITIONS: Apical Periodontitis
Keywords: Apical Patency; Root Canal Treatment
MeSH Terms: conditions — Periapical Periodontitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patency Group (Experimental): apical patency was maintained during chemomechanical preparation
  Interventions: Procedure: Apical patency
- Non Patency Group (No Intervention): Apical patency was not maintained during chemomechanical preparation

INTERVENTIONS:
Procedure: Apical patency — Apical patency was maintained by passing a #10 K file 1 mm beyond working length between every instrument change while doing chemomechanical preparation
  Arms: Patency Group

SUMMARY:
Maintaining Apical patency during root canal treatment is a widely followed methodology in modern endodontic treatment protocols. It involves passing of a small #08 or #10 K file through the apical foramen during root canal shaping without widening it. it is done to keep the foramen and apical thirds of root canal free of debris. proponents of the procedure claim it to improve irrigation; provide better tactile feedback; reduce the chances of procedural errors; reduce transportation and reduce pain following root canal procedures. however, there is no clinical trial which specifically evaluates the effect of apical patency on outcome of root canal procedure. hence this study was designed to evaluate the effect of apical patency on outcome of root canal treatment.

DETAILED DESCRIPTION:
AIM:

1. To assess the role of maintaining Apical Patency on success of primary Non-Surgical Root Canal Treatment (NSRCT) in Non-Vital teeth.
2. To evaluate the incidence of post-operative complications such as pain, flare-up etc with and without maintaining apical patency.

Study subjects were recruited from the pool of patients referred for the initial non-surgical root canal treatment to the post graduate department Of Conservative Dentistry & Endodontics at PGIDS, Rohtak (Haryana). Patients requiring Root Canal Treatment following the diagnosis pulpal necrosis in mature mandibular first molar were selected for the study.

Clinical procedure:

Subjects were randomly allocated to one of the two study groups (patency or non-patency). It was ensured that neither the patient, nor the primary investigator was aware of the treatment protocol before completing the consent process. After administration of local anesthesia, rubber dam isolation of the involved tooth was done. Caries excavation was done and access cavity prepared using carbide burs in high speed handpiece with copious irrigation. Debridement of the pulp chamber was done and all canal orifices identified. Working length was obtained with the help of electronic apex locator (Root ZX) and confirmed radiographically. ProTaper S1 and Sx were used to flare coronal thirds and WL was reconfirmed with apex locator. Hand files No. 10, 15 and 20 were used till working length (WL) to prepare a smooth reproducible glide path. ProTaper S1 and S2 were used till WL, followed by the use of ProTaper finishing files (F1/F2/F3) to prepare the canal to desired size as determined by the operator. Copious irrigation with 3% Sodium Hypochlorite was carried out throughout the procedure with the use of 27-gauge side vented needle.

In patency group, a #10 K- file was passed 1mm beyond the WL between each instrument change, while in non-patency group it was carried till the WL. In patency group, a final radiograph was taken after completion of preparation, with a #10 file placed 1mm beyond the WL to confirm patency.

After enlargement, the canals were irrigated with 5ml 17% EDTA for 1 min followed by irrigation with 5ml 3% NaOCl. Canals were dried with absorbent paper points and filled with a paste made by mixing Calcium hydroxide powder with 2% Chlorhexidine liquid; and the access cavity restored with intermediate restorative material (IRM). The patient was recalled after 1 week. At the next appointment, the paste was removed with H- files and copious irrigation with 3% NaOCl. Canals were examined under operating microscpe. A final rinse of 5ml 17% EDTA and 5ml 3% NaOCl was done and canals dried with paper points. Canals were obturated with the GuttaPercha and Zinc Oxide- Eugenol based sealer. After obturation, the cavity was restored with Silver Amalgam/Composite/Full coverage crown. Immediate post-operative radiograph was then taken using preset exposure parameters with Rinn paralleling device; and processed manually. Follow up clinical and radiographic examination was carried out every 3 months, till a 12 month period.

Data Gathering Details:

Preoperative and intraoperative data were obtained from patient records. Diagnostic and treatment information was meticulously recorded on a custom designed endodontic treatment form by the operator. Diagnostic and treatment details for each patient were extracted from the records by the principal investigator.

Assessment of treatment outcome:

Treatment outcome was judged on the basis of clinical and radiographic findings recorded at the follow up visit and comparison of the radiographs obtained at post obturation and the follow-up visit

Radiographic success:

Change in Periapical Index (PAI) scores (Orstaviket al) observed at 12-months was noted. Scoring of each tooth was done according to the following five point scale (PAI):

PAI Score Description of radiographic findings

1. Normal periapical structures
2. Small changes in bone structure
3. Changes in bone structure with some mineral loss
4. Periodontitis with well-defined radiolucent area
5. Severe periodontitis with exacerbating features

Three experienced observers with no knowledge of the treatment protocol independently examined immediate post obturation and follow-up radiographs, mounted side by side, under controlled conditions. The treatment was considered successful only when both clinical and radiographic criteria were met. In multirooted teeth, the worst outcome by root decided the overall outcome for the tooth. In the event of disagreement, the three observers met to discuss their findings and came to an agreement. In the absence of unanimity, the majority decision was taken.

Clinical Success:

Absence of pain and tenderness to palpation/ percussion, absence of sinus or any associated soft tissue swelling, tooth mobility of grade-I or less, and no deterioration in periodontal probing depth as compared with baseline measurements comprised the criteria for clinical success.

ELIGIBILITY:
Inclusion Criteria:

1. Mature permanent mandibular first molars
2. Diagnosis of pulp necrosis, as confirmed by negative response to cold and electrical tests
3. Radiographic evidence of apical periodontitis (minimum size ≥ 2.0 × 2.0 mm)
4. Probing depth < 4mm

Exclusion Criteria:

1. Non willingness to participate in study
2. younger than 18 years of age
3. Pregnant, diabetic or immunocompromised
4. Prior endodontic treatment of the same tooth
5. History of antibiotic use in past one month or requiring antibiotic pre-medication
6. unrestorable teeth, fractured or perforated roots, grade 3 mobility

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2013-05-01 (Actual); Primary Completion 2013-11-28 (Actual); Study Completion 2014-11-30 (Actual)

PRIMARY OUTCOMES:
Change in periapical radiolucency | Baseline to 12-month
  The change observed in periapical radiolucency at the 12-month follow-up visit was used to assess the success of the treatment

SECONDARY OUTCOMES:
Clinical success | Baseline to 12-month
  Absence of pain and tenderness to percussion/palpation, the absence of sinus or any associated soft-tissue swelling, tooth mobility of grade 1 or less, and no deterioration in periodontal probing depth as compared with baseline measurements